CLINICAL TRIAL: NCT00142584
Title: An Open-label, Randomized Study Evaluating the Long-term Effects of Metoprolol (MET) Versus Nebivolol (NEB) as Monotherapy or in Combination With Amlodipine or Hydrochlorothiazide for the Treatment of Patients With Hypertension
Brief Title: Evaluation of the Long-term Safety and Tolerability of Metoprolol Versus Nebivolol in Patients With Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mylan Bertek Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEB324
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Results first posted 2022-03-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-02

CONDITIONS: Hypertension
Keywords: safety and tolerability study; hypertension; beta-blockers
MeSH Terms: conditions — Hypertension | interventions — Nebivolol; Metoprolol

ARMS (2):
- 1-NEB (Experimental): Nebivolol
  Interventions: Drug: Nebivolol (NEB)
- 2-MET (Active Comparator): Metoprolol
  Interventions: Drug: Metoprolol (MET)

INTERVENTIONS:
Drug: Nebivolol (NEB) — Patients randomized to nebivolol will initiate therapy with nebivolol 5 mg once daily for 4 weeks.
  Arms: 1-NEB
Drug: Metoprolol (MET) — Patients randomized to metoprolol will initiate therapy with 100 mg once daily for 4 weeks.
  Arms: 2-MET

SUMMARY:
The purpose of this study is to evaluate long-term safety,tolerability and blood pressure effects of metoprolol versus nebivolol in patients with hypertension. These drugs may be given alone or in combination with other drugs that are commonly used in the treatment of hypertension

DETAILED DESCRIPTION:
Approximately 50 million Americans have hypertension defined as a systolic blood pressure (SBP) greater then or equal to 140 mmHg and/or a diastolic blood pressure (DBP) greater then or equal to 90 mmHg. To control blood pressure, more than 2 agents are required in many patients. The current study is a randomized, titration-to-effect, open-label, multi center study. Patients will be randomized to either nebivolol or metoprolol. The dose of the randomized treatment can be titrated as needed to achieve blood pressure control. If necessary, additional antihypertensive agents (calcium antagonist, diuretic, etc.) can be added to achieve control. Patients will be seen every 1-3 months for approximately 18 months to assess long-term safety, tolerability and effectiveness of nebivolol versus metoprolol.

ELIGIBILITY:
Inclusion Criteria:

* Completion of previous nebivolol study
* Stage 1-2 Hypertension (HTN) at baseline of first study

Exclusion Criteria:

* Recent myocardial infarction or stroke
* Contraindications to beta blocker therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2005-08; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Betty S Riggs, MD, MBA, Study Director — Mylan Pharmaceuticals Inc
Locations (1):
- Mylan Pharmaceuticals Inc., Morgantown, West Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 1-NEB: Nebivolol
  Nebivolol: Patients randomized to nebivolol will initiate therapy with nebivolol 5 mg once daily for 4 weeks.
- 2-MET: Metoprolol
  Metoprolol: Patients randomized to metoprolol will initiate therapy with 100 mg once daily for 4 weeks.
Period: Overall Study
Arm/Group | 1-NEB | 2-MET
Started | 252 | 84
Completed | 108 | 28
Not Completed | 144 | 56
Not completed — Sponsor Termination of Study, etc. | 72 | 16
Not completed — Withdrawal by Subject | 30 | 16
Not completed — Lost to Follow-up | 22 | 12
Not completed — Adverse Event | 14 | 5
Not completed — Protocol Violation | 4 | 7
Not completed — Treatment Failure | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1-NEB | 2-MET | Total
Number analyzed (Participants) | 252 | 84 | 336
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (9.86) | 50.1 (9.76) | 50.6 (9.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 44 | 174
  Male | 122 | 40 | 162
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 252 | 84 | 336
Region of Enrollment [Number; unit: participants]
  United States | 252 | 84 | 336

OUTCOME MEASURES:

1. Primary Outcome: Change in Average Sitting Diastolic Blood Pressure (DBP) Taken at Trough at the End of Treatment Compared to Baseline
Description: The primary efficacy parameter was the change in the average trough sitting DBP at the end of treatment (Visit 10 or Early Termination) compared with baseline (baseline was defined as the baseline visit in Study NEB 310 [NCT00145210]).
Time Frame: Through study duration (approximately 18 months)
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- 1-NEB: Nebivolol (NEB)
  Nebivolol: Patients randomized to nebivolol will initiate therapy with nebivolol 5 mg once daily for 4 weeks.
- 2-MET: Metoprolol (MET)
  Metoprolol: Patients randomized to metoprolol will initiate therapy with 100 mg once daily for 4 weeks.
Arm/Group | 1-NEB | 2-MET
Number analyzed (Participants) | 252 | 84
mm Hg | -14.0 (9.80) | -10.9 (8.73)

2. Secondary Outcome: Change From Baseline in Mean Trough Sitting Diastolic Blood Pressure (DBP) at Each Study Visit (Visits 1 Through 9) Compared to Baseline
Description: Data for the analysis of the change from baseline in mean trough sitting DBP at each study visit (Visits 1 through 9) compared with baseline (baseline was defined as the baseline visit in Study NEB 310 [NCT00145210]) by treatment group are provided below.
Time Frame: Through study completion (approximately 18 months)
Population: The overall number of participants analyzed equals the number of randomized patients at study start; the numbers analyzed at each visit equal the number of patients at each treatment visit.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | 1-NEB | 2-MET
Number analyzed (Participants) | 252 | 84
mm Hg
  Visit 1 | -8.3 (8.24) | -8.4 (9.15)
  Visit 2: number analyzed (Participants) | 236 | 79
  Visit 2 | -8.4 (8.39) | -8.4 (7.89)
  Visit 3: number analyzed (Participants) | 221 | 76
  Visit 3 | -10.6 (8.51) | -9.8 (8.07)
  Visit 4: number analyzed (Participants) | 212 | 71
  Visit 4 | -12.1 (8.55) | -10.7 (8.20)
  Visit 5: number analyzed (Participants) | 201 | 67
  Visit 5 | -13.0 (8.03) | -12.4 (7.41)
  Visit 6: number analyzed (Participants) | 171 | 56
  Visit 6 | -14.5 (8.49) | -12.1 (7.94)
  Visit 7: number analyzed (Participants) | 150 | 50
  Visit 7 | -15.5 (8.55) | -13.1 (8.74)
  Visit 8: number analyzed (Participants) | 129 | 38
  Visit 8 | -16.3 (8.59) | -12.4 (6.78)
  Visit 9: number analyzed (Participants) | 116 | 34
  Visit 9 | -16.7 (7.91) | -13.7 (7.05)

3. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: Summary of Participants that experienced one or more TEAEs by Treatment Group-Safety Population
Time Frame: Through study completion (approximately 18 months)
Measure: Count of Participants; unit: Participants
Arm/Group | 1-NEB | 2-MET
Number analyzed (Participants) | 252 | 84
Participants | 150 | 51

ADVERSE EVENTS:
Time Frame: Through study completion (approximately 18 months)
Arm/Group | 1-NEB | 2-MET
All-Cause Mortality (participants affected / at risk) | 3/252 | 0/84
Serious Adverse Events (participants affected / at risk) | 11/252 | 2/84
Other Adverse Events (participants affected / at risk) | 74/252 | 28/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1-NEB (N=252) | 2-MET (N=84)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
CHEST PAIN (General disorders) | 1 (1) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0)
ANIMAL BITE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
WOUND (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 2 (2) | 0 (0)
CEREBRAL ARTERY OCCLUSION (Nervous system disorders) | 1 (1) | 0 (0)
CERVICAL MYELOPATHY (Nervous system disorders) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0)
ALCOHOLISM (Psychiatric disorders) | 1 (1) | 0 (0)
CONVERSION DISORDER (Psychiatric disorders) | 1 (1) | 0 (0)
PROSTATITIS (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1-NEB (N=252) | 2-MET (N=84)
HEADACHE (Nervous system disorders) | 17 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 4
Nasopharyngitis (Infections and infestations) | 12 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 4
Upper respiratory tract infection (Infections and infestations) | 8 | 4
Peripheral edema (General disorders) | 7 | 4
Sinusitis (Infections and infestations) | 5 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator Study Agreement: Publication Clause - Details of the Study and its results shall not be publicized or published in any form without prior consent of Covance and the Sponsor, Mylan.